CLINICAL TRIAL: NCT02833090
Title: The Plasma Serotonin and Aortic Stenosis: a Pilot Study.
Acronym: SERAOPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09 238 03
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Other): Control group had biomarkers.
  Interventions: Procedure: biomarkers
- Group 2 (Experimental): Biomarkers
  Interventions: Procedure: biomarkers
- Group 3 (Experimental): Biomarkers
  Interventions: Procedure: biomarkers
- Group 4 (Experimental): Biomarkers
  Interventions: Procedure: biomarkers

INTERVENTIONS:
Procedure: biomarkers — transthoracic echocardiography, radial, and aortic arterial blood sampling

SUMMARY:
The goal of this study is to describe the increase in plasma serotonin or 5-hydroxytryptamine (5-HT) in patient with increased severity of aortic stenosis and increased weight cardiac muscle.

DETAILED DESCRIPTION:
Calcific aortic stenosis is the most frequent valve disease in adults. Without therapeutic strategy, this disease leads to heart failure and death. Surgical aortic valve replacement is now a well tolerated cardiac surgery leading to excellent outcomes. Until recently, calcific aortic stenosis was considered to be histopathologically degenerative or passive in origin. It is now recognized, however, as a complex cellular process with features of atherosclerosis. It has been observed that drugs may slow dawn the progression of aortic stenosis in observational studies.

It has been suggested that serotonin, a monoamine neurotransmitter and a peripheral signal mediator, may be involved in the progression of aortic stenosis and also in its consequences on myocardium hypertrophy.

In the blood, serotonin in mainly stored in platelets, which release serotonin involved in post-injury vasoconstriction, thrombus formation, fibrosis and atherogenesis.

This study hypothesized those patients with aortic stenosis exhibit higher circulating serotonin levels than their counterparts without heart disease. In addition to circulating serotonin, its metabolite 5-HIAA will be systematically measured on all patients.

This study would allow to determine the potential of plasma serotonin as a prognosis marker and perhaps suggest the discovery of new targets for treatment of aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 : non aortic stenosis
* Goup 2, 3 and 4 : aortic stenosis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measurements of 5-HT | baseline
  Measurement of 5-HT were performed by high pressure liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Measurements of acide 5-hydroxy-indol-acetic (5-HIAA) | Baseline
  Measurements of 5-HT monoamine oxidase (MAO)-A-dependent degradation product, 5-HIAA, were performed by HPLC
Arterial platelet activation | Baseline
  Arterial platelet activation was assessed by flow cytometry analysis of platelet surface expression of P-selectin and activated integrin GPIIb/IIIa

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lairez, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rouzaud-Laborde C, Delmas C, Pizzinat N, Tortosa F, Garcia C, Mialet-Perez J, Payrastre B, Sie P, Spreux-Varoquaux O, Sallerin B, Carrie D, Galinier M, Parini A, Lairez O. Platelet activation and arterial peripheral serotonin turnover in cardiac remodeling associated to aortic stenosis. Am J Hematol. 2015 Jan;90(1):15-9. doi: 10.1002/ajh.23855. PMID 25242620